CLINICAL TRIAL: NCT00003212
Title: Randomized Phase III Trial of Two Investigational Schedules of Ifosfamide vs. Standard Dose Doxorubicin in Patients With Advanced or Metastatic Soft Tissue Sarcoma
Brief Title: Ifosfamide or Doxorubicin in Treating Patients With Advanced or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-62971; EORTC-62971
Record Dates: First submitted 1999-11-01; First posted 2004-03-12 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Sarcoma
Keywords: adult angiosarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult neurofibrosarcoma; adult synovial sarcoma; recurrent adult soft tissue sarcoma; adult malignant fibrous histiocytoma; adult malignant hemangiopericytoma; adult rhabdomyosarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant; Rhabdomyosarcoma | interventions — Doxorubicin; Ifosfamide

INTERVENTIONS:
Drug: doxorubicin hydrochloride
Drug: ifosfamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether ifosfamide or doxorubicin is more effective for advanced or metastatic soft tissue sarcoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of ifosfamide with that of doxorubicin in treating patients who have advanced or metastatic soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the progression free survival rate in patients with advanced or metastatic soft tissue sarcoma treated with either of two different regimens of ifosfamide or doxorubicin. II. Assess the toxic effects of these therapies and response rate in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized into one of 3 arms (continuous ifosfamide, ifosfamide daily for 3 days, or doxorubicin). Patients are stratified by performance status (0 vs 1), liver involvement (no vs yes), histological type (leiomyosarcoma vs synovial sarcoma vs other), and histological grade (1 vs 2 vs 3). Arm I: Patients receive doxorubicin by bolus infusion for 5-20 minutes once every 3 weeks. Arm II: Patients receive ifosfamide by intravenous infusion for 4 hours on days 1, 2, and 3 every three weeks. Arm III: Patients receive ifosfamide by intravenous infusion for 72 hours every 3 weeks. Patients are assessed after every 2 courses of therapy. Each course of therapy consists of 3 weeks of treatment. Patients may receive a maximum of 6 courses of therapy in the absence of toxicity and disease progression. Patients are followed every 12 weeks for survival.

PROJECTED ACCRUAL: A total of 780 patients (260 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced or metastatic soft tissue sarcoma including the following: Malignant fibrous histiocytoma Liposarcoma Rhabdomyosarcoma Synovial sarcoma Malignant paraganglioma Fibrosarcoma Leiomyosarcoma Angiosarcoma including haemangiopericytoma Neurogenic sarcoma Unclassified sarcoma Mixed mesodermal tumor of the uterus Measurable disease with evidence of progression in prior 6 weeks No symptomatic or known CNS metastases

PATIENT CHARACTERISTICS: Age: 15 to 65 Performance status: WHO 0-1 Life expectancy: Not specified Hematopoietic: WBC at least 3000/mm3 Neutrophil count greater than 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater 1.75 mg/dL Albumin at least 25 g/L Renal: Creatinine clearance greater than 70 mL/min Cardiovascular: No history of uncontrolled cardiovascular disease Other: Fertile women must use effective contraception No other severe medical illness including psychosis No prior primary malignant tumor except: Adequately treated carcinoma in situ of the cervix Basal cell carcinoma

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No radiotherapy to the sole index lesion Surgery: Not specified

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 1998-01; Primary Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul C. Lorigan, MD, Study Chair — The Christie NHS Foundation Trust
Locations (23):
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Denmark (2):
  - Aarhus Kommunehospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (2):
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Grosshadern, Munich
- National Institute of Oncology, Budapest, Hungary
- Netherlands (4):
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- National Cancer Institute - Bratislava, Bratislava, Slovakia
- Hospital Insular de Gran Canaria, Las Palmas, Spain
- United Kingdom (7):
  - St. James's Hospital, Leeds, England
  - Royal Marsden NHS Trust, London, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Weston Park Hospital, Sheffield, England

REFERENCES:
- [Result] Lorigan P, Verweij J, Papai Z, Rodenhuis S, Le Cesne A, Leahy MG, Radford JA, Van Glabbeke MM, Kirkpatrick A, Hogendoorn PC, Blay JY; European Organisation for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group Study. Phase III trial of two investigational schedules of ifosfamide compared with standard-dose doxorubicin in advanced or metastatic soft tissue sarcoma: a European Organisation for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group Study. J Clin Oncol. 2007 Jul 20;25(21):3144-50. doi: 10.1200/JCO.2006.09.7717. PMID 17634494